CLINICAL TRIAL: NCT06292390
Title: The Effect Of Pet Therapy Applıed To Elderly Indıvıduals Lıvıng In A Nursıng Home On Sleep And Qualıty Of Lıfe
Brief Title: The Effect Of Pet Therapy Applıed To Elders's Sleep And Qualıty Of Lıfe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Cansu Yilmaz, Lecturer, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AIBU-SBF-CY-09
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Pet Therapy Effect of Sleep and Quality of Life
Keywords: poor quality of life; problems of sleeping; sleeplessness; pet therapy; nursing practices
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Animal Assisted Therapy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial (Two groups with intervention and control group)
Who Masked: Investigator, Outcomes Assessor
Masking Description: A pollster who did not know the people in the control and intervention group was selected and collected the data. The SPSS data were entered by someone selected other than the surveyor and the researcher. Thus, the study was conducted as a double-blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Pet therapy was applied to the individuals in the intervention group for 6 weeks in addition to their normal routine lives. This therapy was applied every 20 minutes, 2 days a week. Repeated measurements were made before therapy, at the end of therapy and 4 weeks after the end of therapy. The scales were collected by the questionnaire by face-to-face interview method.
  Interventions: Other: Pet Therapy
- Control Group (No Intervention): The elderly in this group have not been given any treatment, they have received routine nursing home care and necessary treatments if any. The first evaluation of the elderly in the control group, 6.week and 10.the necessary measurements were made with the scales three times a week in total. The scales were collected by the questionnaire by face-to-face interview method.

INTERVENTIONS:
Other: Pet Therapy — Pet therapy was applied to the individuals in the intervention group for 6 weeks in addition to their normal routine lives. This therapy was applied every 20 minutes, 2 days a week. Repeated measurements were made before therapy, at the end of therapy and 4 weeks after the end of therapy.
  Arms: Intervention Group

SUMMARY:
Quality of life is defined as functional abilities that include the ability to fulfill an individual social role, the degree and quality of social interaction, mental health, physical competence, somatic senses such as pain, and satisfaction with life. The World Health Organization (WHO) defined quality of life in 1947 as a decrease not only in disease, disorder or disability, but also in physical, mental and social well-being. Old age is one of the situations in which the quality of life decreases. It is reported that the poor social and financial situation of individuals, low educational level, gender, lack of physical movement, decreased daily life activity level, decreased mobility ability, fall anxiety, sleep problems and other conditions that cause disability are determinants of the quality of life. According to the results of Bloom et al.'s study, elderly people wake up at night due to health problems.

According to the literature, the sleep and life of pet therapy applied to elderly individuals living in a nursing home there have not been any studies examining the effect on quality. For this reason, it was aimed to conduct this study in order to determine the effect of pet therapy applied to elderly individuals living in a nursing home on sleep and quality of life.

The study was planned to be conducted in a randomized controlled manner in order to determine the effect of pet therapy applied for one hour twice a week for 6 weeks to elderly people living in a nursing home in Tokat province on sleep pattern and quality of life. In the study, gender, age group and the presence of chronic diseases were taken as equivalence criteria. Since conducting the study single-blind will increase the reliability of the study, the application of the scales was applied by another researcher/surveyor other than the main researcher.

DETAILED DESCRIPTION:
The study was planned to be conducted in a randomized controlled manner in order to determine the effect of pet therapy applied for one hour twice a week for 6 weeks to elderly people living in a nursing home in Tokat province on sleep pattern and quality of life.

The universe of the research consists of 74 elderly elderly individuals who are located in a nursing home in Tokat province and meet the criteria for inclusion.

As a result of the calculations; the minimum sample volume that will provide the test power (1-β) = 0.95 was calculated as a total of 46 (23 interventions + 23 controls) people, and the net power of this study was determined as 0.952.

In the research, the data will be collected through the 'Elderly Person Introduction Form" CASP-19 Quality of Life Scale and PUKI sleep quality scale and Mini Mental Test (MMT). Since conducting the study double-blind will increase the reliability of the study, the application of the scales was applied by another researcher/surveyor other than the main researcher.

The Control Group Protocol:

The elderly in this group have not been given any treatment, they have received routine nursing home care and necessary treatments if any. The first evaluation of the elderly in the control group, 6.week and 10.the necessary measurements were made with the scales three times a week in total. The scales were collected by the questionnaire by face-to-face interview method.

Intervention Group Protocol:

After the data collection process of the control group was completed, the data collection process of the intervention group and pet therapy were applied. As a result of literature review; there is no clear duration for pet therapy and it was found that the average activity duration was 10-30 minutes, 4-12 weeks and 6-24 sessions. Based on this literature information; for this research, pet therapy pet therapy was applied for a total of 6 weeks and 12 sessions, 2 times a week for an average of 20 minutes for each elderly individual. End of therapy 6.week rating and 10.the scale was applied three times in total, including control measurement after a week of therapy. The scales applied by the animal therapy researcher were collected by the face-to-face interview method by the interviewer who did not know the groups.

In the evaluation of data, IBM SPSS Statistics 25.0 (IBM Corp. Released 2017. IBM SPSS Statistics for Windows, Version 25.0.Armonk, NY: IBM Corp.) the statistical package program was used. The normal distribution of the data of numerical variables was evaluated by Shapiro-Wilk normality test/Kruskal Wallis test and Q-Q graphs. Spearman correlation analysis was performed to determine the relationship between the dimensions. Dec. Statistically, a value of p≤0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Tokat- Living in a nursing home,
* According to expert opinion, elderly people who received a minimum of 24 points in Mini Mental Test assessments,
* Able to communicate,
* Those who are not immobile and able to do activities with a dog,
* Not allergic to a dog,
* Not having a phobia of dogs,
* Sedative / antisedative, insomnia / hypersomnia,
* Elderly who agreed to participate in the study

Exclusion Criteria:

* People who are immobile and unable to do activities with the dog,
* Individuals who cannot communicate,
* (According to expert view)Those who score below 24 points of Mini Mental Test,
* Those who are allergic to dogs,
* Those who have a phobia of dogs,
* Those who use medications that will affect sleep processes, such as sedatives /antisedatives, insomnia/hypersomnia,
* People who do not want to participate in the study.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
PUKI | First week, the end of six week and end of ten week.
  PUKI was developed by Buysse et al. in 1989 and has been shown to have sufficient internal consistency (Cronbach alpha= 0.80), test-retest reliability and validity (Buysse Reynolds Monk Berman and Kupfer 1989). The validity and reliability study of PUKI in our country was conducted by Ağargün et al. In this study, the Cronbach alpha value of the scale was found to be 0.79 (Cronbach alpha= 0.79). The total score has a value between 0-21.Dec. High values indicate that the quality of sleep is poor, the level of sleep disorders is high. A total score above 5 indicates that sleep quality is clinically poor.

SECONDARY OUTCOMES:
CASP-19 QUALITY OF LIFE | First week, the end of six week and end of ten week.
  The CASP-19 scale was developed by Hyde et al. in 2003 to measure the quality of life of elderly people. The scale consists of 19 items. The items of the scale are scored between 0-3 points.Dec. An increase in the total score indicates an increase in the quality of life. As a result of the factor analysis conducted by Hyde et al. for structure validity, it was found that the scale consists of 4 sub-dimensions, the Cronbach's alpha values of each sub-dimension are between 0. Dec.9-Dec.77, the item total score correlation coefficients are between r= 0.35 and r= 0.67.

CONTACTS AND LOCATIONS:
Overall Officials: Cansu YILMAZ, Principal Investigator — https://www.gop.edu.tr/AkademikOzgecmis/6508/cansu-yilmaz; Pınar TEKINSOY KARTIN, Study Director — https://avesis.erciyes.edu.tr/ptekinsoy
Locations (1):
- Nursing Home, Tokat Province, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No